CLINICAL TRIAL: NCT02211846
Title: A Multicentre, Open-label, Single Ascending Dose Phase 1 Study to Evaluate the Pharmacokinetics, Safety and Tolerability of Mirabegron OCAS Tablets in Pediatric Subjects From 5 to Less Than 18 Years of Age With Neurogenic Detrusor Overactivity (NDO) or Overactive Bladder (OAB)
Brief Title: A Study to Evaluate the Pharmacokinetics, Safety and Tolerability of Mirabegron OCAS (Oral Controlled Absorption System) in Pediatric Subjects With Neurogenic Detrusor Overactivity or Overactive Bladder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 178-CL-202; 2014-000340-15 (EudraCT Number)
Record Dates: First submitted 2014-08-06; First posted 2014-08-08 (Estimated); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Neurogenic Detrusor Overactivity; Overactive Bladder; Pharmacokinetics of Mirabegron
Keywords: Pharmacokinetics; Mirabegron; Neurogenic detrusor overactivity (NDO); Overactive bladder (OAB)
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — mirabegron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mirabegron (Experimental): Administered under fed and fasted conditions
  Interventions: Drug: Mirabegron

INTERVENTIONS:
Drug: Mirabegron — oral
  Other Names: Myrbetriq; Betmiga; Betanis

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics as well as the safety and tolerability of mirabegron OCAS tablets after single-dose administration at different dose levels in children and adolescents with NDO or OAB.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a documented diagnosis of:

  * Neurogenic detrusor overactivity (NDO), or
  * Idiopathic overactive bladder (OAB) according to International Children's Continence Society (ICCS) criteria.
* Subject's weight/height:

  * Subject should have a body weight of ≥ 20.0 kg (all cohorts).
  * For NDO: subject is not suffering from malnutrition and is not severely overweight, in the opinion of the Investigator.
  * For OAB: subject's weight and height are within the normal percentiles (3rd to 97th percentile) according to Centers for Disease Control and Prevention (CDC) growth charts.
* Subject is able to swallow the study medication in accordance with the protocol.
* Female subject must either:

  * Be of non-childbearing potential:
  * Clearly pre-menarchal or in the judgment of the Investigator is pre-menarchal
  * Documented surgically sterile.
  * Or, if of childbearing potential: Agree not to try to become pregnant during the study and for 28 days after the final study drug administration,
  * And have a negative urine pregnancy test pre-dose Day 1,
  * And, if heterosexually active agree to consistently use two forms of highly effective form of birth control starting at screening and throughout the study period and for 28 days after the final study drug administration.
* Female subjects must agree not to breastfeed starting at screening and throughout the study period, and for 28 days after the last study drug administration.
* Female subject must not donate ova starting at screening and throughout the study period, and for 28 days after the final study drug administration.
* Male subject and their female spouse/partner who are of childbearing potential must be using a highly effective form of contraception consisting of two forms of birth control (one of which must be a barrier method) starting at screening and continuing throughout the study period, and for 28 days after the final study drug administration.
* Male subject must not donate sperm starting at Screening and throughout the study period, and for 90 days after study drug administration.
* Subject and subject's parent(s)/legal guardian agree that the subject will not participate in another interventional study while on treatment.
* Subject and subject's parent(s)/legal guardian are willing and able to comply with the study requirements and with the concomitant medication restrictions

Exclusion Criteria At Screening:

* Subject is pregnant.
* Subject has a known history of QTc prolongation or risk of QT prolongation (e.g. hypokalemia, family history of Long QT Syndrome).
* Subject has an abnormal (mean) pulse rate according to the ranges specified below: age 5 to less than 8 years: < 60 bpm or > 110 bpm; age 8 to less than 12 years: < 55 bpm or > 100 bpm; age 12 to less than 18 years: < 50 bpm or > 100 bpm.
* Subject has any clinically significant ECG abnormality.
* Subject has mean systolic blood pressure greater than the 95th percentile according to age and height and/or greater than 140 mmHg [National Institute of Health, 2005].
* Subject has any clinically significant or unstable medical condition or disorder which, in the opinion of the Investigator, precludes the subject from participating in the study.
* Subject has aspartate aminotransferase (AST) or alanine aminotransferase (ALT) greater than or equal to 2 times the upper limit of normal (ULN) or total bilirubin greater than or equal to 1.5 times the ULN.
* Subject has severe renal impairment (estimated glomerular filtration rate (MDRD) < 30 mL/min).
* Subject has any other clinically significant out of range results of urinalysis, biochemistry or hematology.
* Subject has a history or current diagnosis of any malignancy.
* Subject has known or suspected hypersensitivity to mirabegron, other ß3-agonists, any of the excipients used in the OCAS tablet formulation or previous severe hypersensitivity to any drug.
* Subject meets any of the contra-indications or precautions for use of mirabegron as mentioned in the Investigator's Brochure (IB).
* Subject has used mirabegron in the past (last intake less than 12 days before planned reference day (Day -4 to Day -1).
* Subject requires ongoing treatment with any of the following prohibited medications:

  * Any anticholinergic/antimuscarinic drugs within 5 half-lives prior to planned reference day (Day -4 to Day -1).
  * Any drugs that are sensitive CYP2D6 substrates with a narrow therapeutic index (such as thioridazine, flecainide, propafenone, imipramine, desipramine) and sensitive P-gp substrates (such as digoxin, dabigatran) within 5 half-lives prior to the planned reference day (Day -4 to Day -1).
  * Any moderate or strong cytochrome CYP3A4/5 or P-gp inhibitors or inducers including natural and herbal remedies (such as itraconazole, rifampicin, phenytoin, carbamazepine, St. John's Wort, grapefruit, Seville orange) within 5 half-lives prior to the planned reference day (Day -4 to Day -1).
* Subject has a positive urinary drug screen test for drugs of abuse.
* Subject donated blood or blood products within 3 months prior to planned Day 1.
* Subject has participated in another clinical trial and/or has taken an investigational drug within 30 days (or 5 half-lives of the investigational drug, whichever is longer) prior to the planned reference day (Day -4 to Day -1).
* Subject's parent(s)/legal guardian is an employee of the Astellas Group, any Contract Research Organization (CRO) involved, or the Investigator site executing the study.
* Subject has current, untreated constipation (or fecal impaction for NDO patients). If the constipation is being consistently treated for the last month, the subject can be included.
* Subject has been administered intradetrusor botulinum toxin injections; except if given > 4 months prior to screening and symptoms reappeared comparable to those before botulinum toxin injections.

Exclusion Criteria At day 1:

* Subject has a positive urinary drug screen test for drugs of abuse.
* Subject has a positive alcohol breath test.
* Subject has used mirabegron in the past (last intake less than 24 days before planned reference day (Day -4 to Day -1).
* Subject requires ongoing treatment with any of the following prohibited medications:

  * Any anticholinergics/antimuscarinics within 5 half-lives prior to intake of the reference day (Day -4 to Day -1).
  * Any drugs that are sensitive CYP2D6 substrates with a narrow therapeutic index (such as thioridazine, flecainide, propafenone, imipramine, desipramine) and sensitive P-gp substrates (such as digoxin, dabigatran) within 5 half-lives prior to the reference day (Day -4 to Day -1).
  * Any moderate or strong cytochrome CYP3A4/5 or P-gp inhibitors or inducers including natural and herbal remedies (such as itraconazole, rifampicin, phenytoin, carbamazepine, St. John's Wort) within 5 half-lives prior to reference day (Day -4 to Day -1).
* Subject donated blood or blood products within 3 months prior to Day 1.
* Subject (female subjects of childbearing potential) has a positive urinary pregnancy test.
* Subject has a current symptomatic urinary tract infection.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2014-09-21 (Actual); Primary Completion 2015-09-21 (Actual); Study Completion 2015-09-21 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter of mirabegron: Cmax | Day 1-7
  Maximum concentration (Cmax)
Pharmacokinetic parameter of mirabegron: tmax | Day 1-7
  The time after dosing when Cmax occurs (tmax)
Pharmacokinetic parameter of mirabegron: AUCinf | Day 1-7
  Area under the curve extrapolated until time is infinity (AUCinf)
Pharmacokinetic parameter of mirabegron: t1/2 | Day 1-7
  Apparent terminal elimination half-life (t1/2 )

SECONDARY OUTCOMES:
Safety as assessed by adverse events, clinical laboratory evaluations, vital signs (including 24-h Holter for heart rate), electrocardiogram (ECG), physical examination, post-void residual volume (PVR) | up to Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Research Physician, Study Director — Astellas Global Development
Locations (13):
- Belgium (4):
  - Site BE32009 Univ.Ziekenhuis Antwerpen, Edegem
  - Site BE32003 Gent University Hospital, Ghent
  - Site BE32004 AZ Groeninge, Campus Vercruyss, Kortrijk
  - Site BE32011 U.Z. Leuven, Leuven
- Denmark (5):
  - Site DK45003 Aalborg Sygehus Nord, Aalborg
  - Site DK45001 Uni Hosp of Aarhus, Skejby, Aarhus
  - Site DK45005 Rigshospitalet, Copenhagen
  - Site DK45004 Børnelægen i Køge, Koege
  - Site DK45002 Kolding Sygehus, Kolding
- Site NO47001 Haukeland Sykehus, Bergen, Norway
- Poland (2):
  - Site PL48003 Uniwersyteckie Centrum Kliniczne, Gdansk
  - Site PL48001 Pomnik-Centrum Zdrowia Dziecka, Warsaw
- Site RS38010 Mother and Child Health Care, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website. — https://astellasclinicalstudyresults.com/patientStudySearch.aspx?RID=;;;178-CL-202